CLINICAL TRIAL: NCT00424177
Title: An Open-label Repeat Dosing Study of Eltrombopag Olamine (SB-497115-GR) in Adult Subjects, With Chronic Idiopathic Thrombocytopenic Purpura (ITP)
Brief Title: Repeated Exposure to Eltrombopag in Adults With Idiopathic Thrombocytopenic Purpura (REPEAT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRA108057
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2012-05

CONDITIONS: Purpura, Thrombocytopaenic, Idiopathic
Keywords: idiopathic thrombocytopenic purpura; ITP; thrombocytopenia; platelets
MeSH Terms: conditions — Purpura; Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- eltrombopag (Experimental)
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — experimental

SUMMARY:
This open-label, repeat dosing study, TRA108057, will evaluate the efficacy, safety and tolerability of eltrombopag, when administered in a repeat, cyclic dosing schedule. The study will describe the effect of repeated (3 cycles), intermittent dosing of eltrombopag on the pharmacodynamics and durability of eltrombopag response as measured by the peripheral platelet counts.

For more information or to see if you qualify, please visit: http://www.itpstudy.com/gov

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

* Subject has signed and dated a written inform consent.
* Adults (≥18 years) diagnosed with chronic ITP according to the American Society of Hematology/British Committee for Standards in Hematology guidelines, and a platelet count between ≥20 Gi/L and ≤50 Gi/L on Day 1 (or within 24 hours prior to dosing on Day 1). In addition, a peripheral blood smear should support the diagnosis of ITP with no evidence of other causes of thrombocytopenia (e.g. pseudothrombocytopenia, myelodysplasia). The physical examination should not suggest any disease which may cause thrombocytopenia other than ITP.
* Subjects who have previously received one or more prior ITP therapies. Previous treatments for ITP include but are not limited to corticosteroids, immunoglobulins, azathioprine, danazol, cyclophosphamide and/or rituximab.
* Subjects must have either initially responded (platelet count >100 Gi/L) to a previous ITP therapy or have had a bone marrow biopsy consistent with ITP within 3 years to rule out myelodysplastic syndromes or other causes of thrombocytopenia.
* It is important to clearly differentiate the effect of eltrombopag on platelet count from the treatment effects of prior and concomitant ITP therapies. Therefore:

  1. Previous therapy for ITP with immunoglobulins (IVIg and anti-D) must have been completed at least 1 week prior to randomization and the platelet count must show a clear downward trend after the last treatment with immunoglobulins. Previous treatment for ITP with splenectomy, rituximab and cyclophosphamide must have been completed at least 4 weeks prior to randomization, or clearly be ineffective.
  2. Subjects treated with concomitant ITP medication (e.g. corticosteroids or azathioprine) must be receiving a dose that has been stable for a least 4 weeks prior to randomization. Subjects treated with cyclosporine A, mycophenolate mofetil or danazol must be receiving a dose that has been stable for at least 3 months prior to randomization.
* Prothrombin time and activated partial thromboplastin time must be within 80 to 120% of normal range with no history of hypercoagulable state.
* A complete blood count (CBC), within the reference range (including differential not indicative of a disorder other than ITP), with the following exceptions:
* Platelet count between ≥20 Gi/L and ≤50 Gi/L on Day 1 (or within 24 hours of Day 1) is required for inclusion.
* Hemoglobin: Subjects with hemoglobin levels between 10g/dL (100g/L) and the lower limit of normal are eligible for inclusion, if anemia is clearly attributable to ITP (excessive blood loss).
* Absolute Neutrophil Count (ANC ) >1500/mL (1.5 x 10^9/L) is required for inclusion (elevated White Blood Cells/ANC above the reference range due to steroid treatment is acceptable).
* The following clinical chemistries MUST NOT exceed the normal reference range by more than 20%: creatinine, Alanine aminotransferase, Aspartate aminotransferase, total bilirubin, total albumin and alkaline phosphatase.
* Subject is practicing an acceptable method of contraception (documented in chart). Female subjects (or female partners of male subjects) must either be of non-childbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal >1 year), or of childbearing potential and use of one of the following acceptable methods of contraception from two weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study:

Complete abstinence from intercourse; Intrauterine device (IUD); Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide); Male partner is sterile prior to entry into the study and is the only partner of the female; Systemic contraceptives (combined or progesterone only).

* Subject is able to understand and comply with protocol requirements and instructions and intends to complete the study as planned.

Exclusion Criteria:

A subject will NOT be eligible for inclusion in this study if any of the following criteria apply:

* Any clinically relevant abnormality, other than ITP, identified on the screening examination or any other medical condition or circumstance, which in the opinion of the investigator makes the subject unsuitable for participation in the study or suggests another primary diagnosis (e.g., thrombocytopenia is secondary to another disease).
* Concurrent malignant disease and/or history of cancer treatment with cytotoxic chemotherapy and/or radiotherapy.
* Any prior history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), AND ≥ two of the following risk factors: hormone replacement therapy, systemic contraception (containing estrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, Antithrombin III deficiency, etc), or any other family history of arterial or venous thrombosis.
* Pre-existing cardiovascular disease (congestive heart failure, New York Heart Association Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a QTc >450 msec.
* Female subjects who are nursing or pregnant (positive serum or urine b-human chorionic gonadotrophin pregnancy test) at screening or pre-dose on Day 1.
* History of alcohol/drug abuse.
* Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
* Subject treated with drugs that affect platelet function (including but not limited to aspirin, clopidogrel and/or Non Steroidal Anti Inflammatory Drugs) or anti-coagulants for > 3 consecutive days within 2 weeks of the study start and until the end of the study.
* History of platelet agglutination abnormality that prevents reliable measurement of platelet counts.
* All subjects with secondary immune thrombocytopenia, including those with laboratory or clinical evidence of human immunodeficiency virus (HIV) infection, anti-phospholipid antibody syndrome, chronic hepatitis B infection, hepatitis C virus infection, or any evidence for active hepatitis at the time of subject screening. If a potential subject has no clinical history that would support HIV infection or hepatitis infection, no further laboratory screening is necessary; however, standard medical practice would suggest further evaluation of patients who have risk factors for these infections.
* Previous participation in a clinical study with eltrombopag.
* Subjects planning to have cataract surgery.
* In France, a subject is neither affiliated with nor a beneficiary of a social security category.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Germany (2):
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Moscow, Russia

REFERENCES:
- [Background] Bussel JB, Saleh MN, Vasey SY, Mayer B, Arning M, Stone NL. Repeated short-term use of eltrombopag in patients with chronic immune thrombocytopenia (ITP). Br J Haematol. 2013 Feb;160(4):538-46. doi: 10.1111/bjh.12169. Epub 2012 Dec 24. PMID 23278590
- [Background] This study has not been published in the scientific literature.
- [Background] Tarantino MD, Fogarty P, Mayer B, Vasey SY, Brainsky A. Efficacy of eltrombopag in management of bleeding symptoms associated with chronic immune thrombocytopenia. Blood Coagul Fibrinolysis. 2013 Apr;24(3):284-96. doi: 10.1097/MBC.0b013e32835fac99. PMID 23492914

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Period: Three cycles of treatment. A cycle is defined as an on-therapy period of up to 6 weeks and an off-therapy period of up to 4 weeks.
Period: Cycle 1: Eltrombopag 50 mg Starting Dose
Arm/Group | Treatment Period
Started | 66
Completed | 55
Not Completed | 11
Not completed — Lack of Efficacy | 8
Not completed — Adverse Event | 1
Not completed — Prolonged Response | 1
Not completed — Relocation | 1
Period: Cycle 2: Eltrombopag 50 or 75 mg
Arm/Group | Treatment Period
Started | 55
Completed | 51
Not Completed | 4
Not completed — Lack of Efficacy | 2
Not completed — Prolonged Response | 1
Not completed — Withdrawal by Subject | 1
Period: Cycle 3: Eltrombopag 50 or 75 mg
Arm/Group | Treatment Period
Started | 51
Completed | 48
Not Completed | 3
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: Male and female participants greater than or equal to 18 years of age with previously treated chronic ITP, as defined according to the American Society of Hematology/British Committee for Standards in Hematology guidelines, who had platelet counts between greater than or equal to 20 gi/L and less than or equal to 50 Gi/L, on the Day 1 visit (or within 24 hours prior to dosing on Day 1).
Arm/Group | Overall Study Population
Number analyzed (Participants) | 66
Age Continuous [Mean (Standard Deviation); unit: years] | 49.6 (14.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 21
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European | 47
  Asian - East Asian | 10
  White - Arabic/North African | 6
  African American/African | 2
  American Indian or Alaska Native | 1
Baseline Platelet Count [Number; unit: participants] — Baseline Platelet Count
  participants
    Less than 20 giga per liter (Gi/L) | 4
    20 Gi/L to 30 Gi/L | 29
    Greater than 30 Gi/L to 50 Gi/L | 31
    Greater than 50 Gi/L | 2
Baseline Splenectomy Status [Number; unit: participants]
  Yes | 20
  No | 46
Use of Idiopathic Thrombocytopenic Purpura Medication at Baseline [Number; unit: participants] — Baseline Idiopathic Thrombocytopenic Purpura (ITP) Medication Use
  participants
    Yes | 22
    No | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Responded (Platelet Count >=50 Gi/L and >=2x Baseline) to Eltrombopag Treatment in Cycle 2 or Cycle 3 Given Participants Responded in Cycle 1
Description: Complete blood count, platelet count by blood draw
Time Frame: Day 42 of each cycle
Population: Primary Analysis Population: All participants who entered the study, received at least 1 dose of eltrombopag, and responded in Cycle 1
Measure: Number; unit: participants
Groups:
- Cycle 1: Eltrombopag 50 mg starting dose. Participants whose platelet count was below 50 Gi/L were permitted to increase to eltrombopag 75 mg on or after Day 22.
- Cycle 2: Same dose of eltrombopag at which participants completed Cycle 1 (eltrombopag 50 or 75 mg)
- Cycle 3: Same dose of eltrombopag at which participants completed Cycle 2 (eltrombopag 50 or 75 mg)
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3
Number analyzed (Participants) | 52 | 51 | 49
participants
  Responders | 52 | 41 | 38
  Non-responders | 0 | 10 | 11
Statistical Analysis 1: Comparison: Cycle 2 vs Cycle 3; Test type: Superiority or Other; Proportion of subjects in Cycle 2 or 3 = 0.87, 95% CI [0.74 to 0.94]

2. Secondary Outcome: Number of Participants Who Responded (Platelet Count Greater Than or Equal to 50 Gi/L and at Least 2x Baseline) for at Least 80 Percent of Their On-therapy Assessments During Weeks 2-6.
Description: CBC, platelet counts
Time Frame: Up to 42 days of dosing
Population: Cycle 1 responders
Measure: Number; unit: participants
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3
Number analyzed (Participants) | 48 | 45 | 43
participants
  At least 80 percent of assessments met criteria | 38 | 35 | 30
  Less than 80 percent of assessments met criteria | 10 | 10 | 13

3. Secondary Outcome: Changes in Participants' Platelet Counts During 3 Cycles of Treatment
Description: Changes from baseline, during on-therapy periods of a cycle, during off-therapy periods of a cycle, and within 4 weeks of permanent discontinuation of eltrombopag treatment.
Time Frame: Up to 1 year
Population: Intent-to-Treat (ITT) Population: All participants who were dispensed study medication
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3
Number analyzed (Participants) | 52 | 52 | 49
Gi/L
  Baseline platelet count | 33.0 [7.0 to 82.0] | 25.0 [0 to 66.0] | 26.0 [8.0 to 167.0]
  Highest on-therapy platelet count | 200.5 [52.0 to 762.0] | 196.0 [31.0 to 613.0] | 174.0 [10.0 to 366.0]
  Lowest on-therapy platelet count | 72.0 [6.0 to 354.0] | 67.5 [7.0 to 454.0] | 59.0 [2.0 to 344.0]
  Highest off-therapy platelet count | 118.5 [0 to 662.0] | 92.5 [12.0 to 701.0] | 125.0 [21.0 to 594.0]
  Lowest off-therapy platelet count | 21.0 [0 to 59.0] | 22.5 [8.0 to 75.0] | 22.0 [0 to 187.0]

4. Secondary Outcome: Number of Participants Who Required Rescue Medication
Description: New idiopathic thrombocytopenic purpura (ITP) medication, increase dose of a concomitant ITP medication from baseline, platelet transfusion, and/or splenectomy
Time Frame: Up to 3 cycles of treatment including follow-up visits following last dose of eltrombopag
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3
Number analyzed (Participants) | 66 | 55 | 51
participants
  Participants who required rescue treatment | 2 | 2 | 10
  Participants who did not require rescue treatment | 64 | 53 | 41

5. Secondary Outcome: Change in Participants Anti-platelet Antibody Levels From Baseline Through Follow-up
Description: Change in participants' anti-platelet antibody levels was measured as the number of samples positive for at least 1 glycoprotein from baseline to follow-up. Serum glycoprotein-specific antigens: GPIIb/IIIa, Ib/IX, and Ia/IIa
Time Frame: Up to 1 year
Population: Safety Population: any participant who received at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Overall Study
Number analyzed (Participants) | 64
participants
  Baseline | 12
  Cycle 2 on-therapy | 6
  Cycle 3 on-therapy | 7
  4-week follow-up | 8
  3-month follow-up | 1
  6-month follow-up | 3

6. Secondary Outcome: Number of Participants With the Indicated Bleeding Signs and Symptoms Using the World Health Organization Bleeding Scale
Description: World health Organization (WHO) Bleeding Scale Grade 0 = no bleeding, Grade 1 = petechiae, Grade 2 = mild blood loss, Grade 3 = gross blood loss, Grade 4 = debilitating blood loss.
Time Frame: Baseline, on-treatment visits (Weeks 1-6), off-treatment visits (Weeks 1-4)
Population: Participants who responded in Cycle 1
Measure: Number; unit: participants
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3
Number analyzed (Participants) | 52 | 52 | 49
participants
  On-therapy, Week 0 (Day 1), n | 52 | 52 | 49
  On-therapy, Week 0, Grade 0 | 26 | 21 | 32
  On-therapy, Week 0, Grades 1-4 | 26 | 31 | 17
  On-therapy, Week 0, Grades 2-4 | 10 | 10 | 6
  On-therapy, Week 1 (Day 8), n | 51 | 51 | 49
  On-therapy, Week 1, Grade 0 | 34 | 36 | 37
  On-therapy, Week 1, Grades 1-4 | 17 | 15 | 12
  On-therapy, Week 1, Grades 2-4 | 4 | 2 | 3
  On-therapy, Week 2 (Day 15), n | 47 | 45 | 43
  On-therapy, Week 2, Grade 0 | 35 | 38 | 32
  On-therapy, Week 2, Grades 1-4 | 12 | 7 | 11
  On-therapy, Week 2, Grades 2-4 | 4 | 2 | 4
  On-therapy, Week 3 (Day 22), n | 33 | 32 | 33
  On-therapy, Week 3, Grade 0 | 28 | 25 | 26
  On-therapy, Week 3, Grades 1-4 | 5 | 7 | 7
  On-therapy, Week 3, Grades 2-4 | 3 | 2 | 2
  On-therapy, Week 4 (Day 29), n | 31 | 28 | 29
  On-therapy, Week 4, Grade 0 | 23 | 22 | 24
  On-therapy, Week 4, Grade 1-4 | 8 | 6 | 5
  On-therapy, Week 4, Grade 2-4 | 2 | 2 | 0
  On-therapy, Week 5 (Day 36), n | 28 | 26 | 29
  On-therapy, Week 5, Grade 0 | 24 | 20 | 24
  On-therapy, Week 5, Grades 1-4 | 4 | 6 | 5
  On-therapy, Week 5, Grades 2-4 | 1 | 3 | 1
  On-therapy, Week 6 (Day 43), n | 25 | 26 | 27
  On-therapy, Week 6, Grade 0 | 22 | 22 | 22
  On-therapy, Week 6, Grades 1-4 | 3 | 4 | 5
  On-therapy, Week 6, Grades 2-4 | 0 | 4 | 1
  Off-therapy, Week 1 (Day 8), n | 47 | 45 | 46
  Off-therapy, Week 1, Grade 0 | 37 | 35 | 42
  Off-therapy, Week 1, Grades 1-4 | 10 | 10 | 4
  Off-therapy, Week 1, Grades 2-4 | 4 | 4 | 0
  Off-therapy, Week 2 (Day 15), n | 37 | 35 | 45
  Off-therapy, Week 2, Grade 0 | 26 | 25 | 30
  Off-therapy, Week 2, Grades 1-4 | 11 | 10 | 15
  Off-therapy, Week 2, Grades 2-4 | 2 | 3 | 2
  Off-therapy, Week 3 (Day 22), n | 28 | 30 | 46
  Off-therapy, Week 3, Grade 0 | 18 | 19 | 30
  Off-therapy, Week 3, Grades 1-4 | 10 | 11 | 16
  Off-therapy, Week 3, Grades 2-4 | 2 | 4 | 7
  Off-therapy, Week 4 (Day 29), n | 7 | 12 | 48
  Off-therapy, Week 4, Grade 0 | 5 | 9 | 30
  Off-therapy, Week 4, Grades 1-4 | 2 | 3 | 18
  Off-therapy, Week 4, Grades 2-4 | 1 | 2 | 6

7. Secondary Outcome: Number of Participants With the Indicated Bleeding Signs and Symptoms Using the ITP Bleeding Score
Description: ITP Bleeding Score: Grade 0 = no bleeding, Grade 1 = mild bleeding, Grade 2 = severe bleeding
Time Frame: Baseline, on-treatment visits (Weeks 1-6), off-treatment visits (Weeks 1-4)
Population: Participants who responded in Cycle 1
Measure: Number; unit: participants
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3
Number analyzed (Participants) | 52 | 52 | 49
participants
  Skin, petechiae, on-therapy, Week 0 (Day 1), n | 50 | 52 | 49
  Skin, petechiae, on-therapy, Week 0, Grade 0 | 35 | 35 | 39
  Skin, petechiae, on-therapy, Week 0, Grade 1 | 14 | 17 | 10
  Skin, petechiae, on-therapy, Week 0, Grade 2 | 1 | 0 | 0
  Skin, petechiae, on-therapy, Week 1 (Day 8), n | 51 | 51 | 48
  Skin, petechiae, on-therapy, Week 1, Grade 0 | 41 | 46 | 44
  Skin, petechiae, on-therapy, Week 1, Grade 1 | 10 | 3 | 3
  Skin, petechiae, on-therapy, Week 1, Grade 2 | 0 | 2 | 1
  Skin, petechiae, on-therapy, Week 2 (Day 15), n | 47 | 45 | 42
  Skin, petechiae, on-therapy, Week 2, Grade 0 | 40 | 43 | 39
  Skin, petechiae, on-therapy, Week 2, Grade 1 | 7 | 2 | 2
  Skin, petechiae, on-therapy, Week 2, Grade 2 | 0 | 0 | 1
  Skin, petechiae, on-therapy, Week 3 (Day 22), n | 33 | 32 | 33
  Skin, petechiae, on-therapy, Week 3, Grade 0 | 31 | 28 | 32
  Skin, petechiae, on-therapy, Week 3, Grade 1 | 2 | 4 | 1
  Skin, petechiae, on-therapy, Week 3, Grade 2 | 0 | 0 | 0
  Skin, petechiae, on-therapy, Week 4 (Day 29), n | 31 | 28 | 29
  Skin, petechiae, on-therapy, Week 4, Grade 0 | 30 | 24 | 28
  Skin, petechiae, on-therapy, Week 4, Grade 1 | 1 | 4 | 1
  Skin, petechiae, on-therapy, Week 4, Grade 2 | 0 | 0 | 0
  Skin, petechiae, on-therapy, Week 5 (Day 36), n | 28 | 26 | 29
  Skin, petechiae, on-therapy, Week 5, Grade 0 | 27 | 21 | 29
  Skin, petechiae, on-therapy, Week 5, Grade 1 | 1 | 5 | 0
  Skin, petechiae, on-therapy, Week 5, Grade 2 | 0 | 0 | 0
  Skin, petechiae, on-therapy, Week 6 (Day 43), n | 24 | 25 | 27
  Skin, petechiae, on-therapy, Week 6, Grade 0 | 24 | 23 | 27
  Skin, petechiae, on-therapy, Week 6, Grade 1 | 0 | 2 | 0
  Skin, petechiae, on-therapy, Week 6, Grade 2 | 0 | 0 | 0
  Skin, petechiae, off-therapy, Week 1 (Day 8), n | 47 | 45 | 48
  Skin, petechiae, off-therapy, Week 1, Grade 0 | 45 | 39 | 45
  Skin, petechiae, off-therapy, Week 1, Grade 1 | 2 | 6 | 3
  Skin, petechiae, off-therapy, Week 1, Grade 2 | 0 | 0 | 0
  Skin, petechiae, off-therapy, Week 2 (Day 15), n | 36 | 35 | 45
  Skin, petechiae, off-therapy, Week 2, Grade 0 | 31 | 30 | 40
  Skin, petechiae, off-therapy, Week 2, Grade 1 | 5 | 5 | 4
  Skin, petechiae, off-therapy, Week 2, Grade 2 | 0 | 0 | 1
  Skin, petechiae, off-therapy, Week 3 (Day 22), n | 29 | 30 | 46
  Skin, petechiae, off-therapy, Week 3, Grade 0 | 27 | 26 | 39
  Skin, petechiae, off-therapy, Week 3, Grade 1 | 2 | 4 | 7
  Skin, petechiae, off-therapy, Week 3, Grade 2 | 0 | 0 | 0
  Skin, petechiae, off-therapy, Week 4 (Day 29), n | 7 | 12 | 48
  Skin, petechiae, off-therapy, Week 4, Grade 0 | 7 | 12 | 41
  Skin, petechiae, off-therapy, Week 4, Grade 1 | 0 | 0 | 6
  Skin, petechiae, off-therapy, Week 4, Grade 2 | 0 | 0 | 1
  Skin, ecchymosis, on-therapy, Week 0 (Day 1), n | 50 | 52 | 49
  Skin, ecchymosis, on-therapy, Week 0, Grade 0 | 31 | 27 | 36
  Skin, ecchymosis, on-therapy, Week 0, Grade 1 | 16 | 25 | 12
  Skin, ecchymosis, on-therapy, Week 0, Grade 2 | 3 | 0 | 1
  Skin, ecchymosis, on-therapy, Week 1 (Day 8), n | 51 | 51 | 48
  Skin, ecchymosis, on-therapy, Week 1, Grade 0 | 39 | 37 | 35
  Skin, ecchymosis, on-therapy, Week 1, Grade 1 | 11 | 13 | 12
  Skin, ecchymosis, on-therapy, Week 1, Grade 2 | 1 | 1 | 1
  Skin, ecchymosis, on-therapy, Week 2 (Day 15), n | 47 | 45 | 42
  Skin, ecchymosis, on-therapy, Week 2, Grade 0 | 42 | 38 | 32
  Skin, ecchymosis, on-therapy, Week 2, Grade 1 | 5 | 7 | 9
  Skin, ecchymosis, on-therapy, Week 2, Grade 2 | 0 | 0 | 1
  Skin, ecchymosis, on-therapy, Week 3 (Day 22), n | 33 | 32 | 33
  Skin, ecchymosis, on-therapy, Week 3, Grade 0 | 28 | 24 | 29
  Skin, ecchymosis, on-therapy, Week 3, Grade 1 | 5 | 8 | 4
  Skin, ecchymosis, on-therapy, Week 3, Grade 2 | 0 | 0 | 0
  Skin, ecchymosis, on-therapy, Week 4 (Day 29), n | 31 | 28 | 29
  Skin, ecchymosis, on-therapy, Week 4, Grade 0 | 24 | 24 | 25
  Skin, ecchymosis, on-therapy, Week 4, Grade 1 | 7 | 4 | 4
  Skin, ecchymosis, on-therapy, Week 4, Grade 2 | 0 | 0 | 0
  Skin, ecchymosis, on-therapy, Week 5 (Day 36), n | 28 | 26 | 29
  Skin, ecchymosis, on-therapy, Week 5, Grade 0 | 25 | 23 | 25
  Skin, ecchymosis, on-therapy, Week 5, Grade 1 | 3 | 3 | 4
  Skin, ecchymosis, on-therapy, Week 5, Grade 2 | 0 | 0 | 0
  Skin, ecchymosis, on-therapy, Week 6 (Day 43), n | 24 | 25 | 27
  Skin, ecchymosis, on-therapy, Week 6, Grade 0 | 20 | 22 | 25
  Skin, ecchymosis, on-therapy, Week 6, Grade 1 | 4 | 3 | 2
  Skin, ecchymosis, on-therapy, Week 6, Grade 2 | 0 | 0 | 0
  Skin, ecchymosis, off-therapy, Week 1 (Day 1), n | 47 | 45 | 48
  Skin, ecchymosis, off-therapy, Week 1, Grade 0 | 42 | 38 | 43
  Skin, ecchymosis, off-therapy, Week 1, Grade 1 | 5 | 7 | 5
  Skin, ecchymosis, off-therapy, Week 1, Grade 2 | 0 | 0 | 0
  Skin, ecchymosis, off-therapy, Week 2 (Day 15), n | 36 | 35 | 45
  Skin, ecchymosis, off-therapy, Week 2, Grade 0 | 26 | 24 | 36
  Skin, ecchymosis, off-therapy, Week 2, Grade 1 | 9 | 11 | 9
  Skin, ecchymosis, off-therapy, Week 2, Grade 2 | 1 | 0 | 0
  Skin, ecchymosis, off-therapy, Week 3 (Day 22), n | 29 | 30 | 46
  Skin, ecchymosis, off-therapy, Week 3, Grade 0 | 16 | 20 | 31
  Skin, ecchymosis, off-therapy, Week 3, Grade 1 | 11 | 9 | 13
  Skin, ecchymosis, off-therapy, Week 3, Grade 2 | 2 | 1 | 2
  Skin, ecchymosis, off-therapy, Week 4 (Day 29), n | 7 | 12 | 48
  Skin, ecchymosis, off-therapy, Week 4, Grade 0 | 6 | 9 | 31
  Skin, ecchymosis, off-therapy, Week 4, Grade 1 | 0 | 3 | 15
  Skin, ecchymosis, off-therapy, Week 4, Grade 2 | 1 | 0 | 2
  Oral, on-therapy, Week 0 (Day 1), n | 50 | 52 | 49
  Oral, on-therapy, Week 0, Grade 0 | 46 | 46 | 46
  Oral, on-therapy, Week 0, Grade 1 | 4 | 5 | 3
  Oral, on-therapy, Week 0, Grade 2 | 0 | 1 | 0
  Oral, on-therapy, Week 1 (Day 8), n | 51 | 51 | 48
  Oral, on-therapy, Week 1, Grade 0 | 49 | 49 | 46
  Oral, on-therapy, Week 1, Grade 1 | 2 | 2 | 2
  Oral, on-therapy, Week 1, Grade 2 | 0 | 0 | 0
  Oral, on-therapy, Week 2 (Day 15), n | 47 | 45 | 42
  Oral, on-therapy, Week 2, Grade 0 | 46 | 43 | 41
  Oral, on-therapy, Week 2, Grade 1 | 1 | 2 | 1
  Oral, on-therapy, Week 2, Grade 2 | 0 | 0 | 0
  Oral, on-therapy, Week 3 (Day 22), n | 33 | 32 | 33
  Oral, on-therapy, Week 3, Grade 0 | 33 | 30 | 31
  Oral, on-therapy, Week 3, Grade 1 | 0 | 2 | 2
  Oral, on-therapy, Week 3, Grade 2 | 0 | 0 | 0
  Oral, on-therapy, Week 4 (Day 29), n | 31 | 28 | 29
  Oral, on-therapy, Week 4, Grade 0 | 30 | 26 | 29
  Oral, on-therapy, Week 4, Grade 1 | 1 | 2 | 0
  Oral, on-therapy, Week 4, Grade 2 | 0 | 0 | 0
  Oral, on-therapy, Week 5 (Day 36), n | 28 | 26 | 29
  Oral, on-therapy, Week 5, Grade 0 | 27 | 24 | 29
  Oral, on-therapy, Week 5, Grade 1 | 1 | 2 | 0
  Oral, on-therapy, Week 5, Grade 2 | 0 | 0 | 0
  Oral, on-therapy, Week 6 (Day 43), n | 24 | 25 | 27
  Oral, on-therapy, Week 6, Grade 0 | 23 | 23 | 26
  Oral, on-therapy, Week 6, Grade 1 | 1 | 2 | 1
  Oral, on-therapy, Week 6, Grade 2 | 0 | 0 | 0
  Oral, off-therapy, Week 1 (Day 8), n | 47 | 45 | 48
  Oral, off-therapy, Week 1, Grade 0 | 45 | 43 | 48
  Oral, off-therapy, Week 1, Grade 1 | 2 | 2 | 0
  Oral, off-therapy, Week 1, Grade 2 | 0 | 0 | 0
  Oral, off-therapy, Week 2 (Day 15), n | 36 | 35 | 45
  Oral, off-therapy, Week 2, Grade 0 | 36 | 35 | 45
  Oral, off-therapy, Week 2, Grade 1 | 0 | 3 | 3
  Oral, off-therapy, Week 2, Grade 2 | 0 | 0 | 0
  Oral, off-therapy, Week 3 (Day 22), n | 29 | 30 | 46
  Oral, off-therapy, Week 3, Grade 0 | 27 | 29 | 41
  Oral, off-therapy, Week 3, Grade 1 | 2 | 1 | 5
  Oral, off-therapy, Week 3, Grade 2 | 0 | 0 | 0
  Oral, off-therapy, Week 4 (Day 29), n | 7 | 12 | 48
  Oral, off-therapy, Week 4, Grade 0 | 7 | 10 | 45
  Oral, off-therapy, Week 4, Grade 1 | 0 | 2 | 2
  Oral, off-therapy, Week 4, Grade 2 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Cycle 1; Cycle 2; Cycle 3: Participants received once-daily treatment for up to 6 weeks, followed by up to 4 weeks off-therapy
- More Than 1 to 30 Days After Last Dose: Adverse events >1 to 30 days after last dose (Post-therapy)
- More Than 30 Days After Last Dose: Adverse events >30 days after last dose (Post-therapy)
- All Cycles: Participants who reported an AE anytime during 3 cycles of treatment. A cycle consisted of once-daily treatment for up to 6 weeks, followed by up to 4 weeks off-therapy.
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3 | More Than 1 to 30 Days After Last Dose | More Than 30 Days After Last Dose | All Cycles
Serious Adverse Events (participants affected / at risk) | 0/66 | 1/55 | 0/51 | 1/66 | 1/66 | 4/66
Other Adverse Events (participants affected / at risk) | 39/66 | 30/55 | 38/51 | 17/66 | 7/66 | 55/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 1 (N=66) | Cycle 2 (N=55) | Cycle 3 (N=51) | More Than 1 to 30 Days After Last Dose (N=66) | More Than 30 Days After Last Dose (N=66) | All Cycles (N=66)
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Ear hemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
Mouth Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cycle 1 (N=66) | Cycle 2 (N=55) | Cycle 3 (N=51) | More Than 1 to 30 Days After Last Dose (N=66) | More Than 30 Days After Last Dose (N=66) | All Cycles (N=66)
Nasopharyngitis (Infections and infestations) | 5 | 2 | 5 | 3 | 1 | 10
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3 | 3 | 0 | 5
Sinusitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 4
Gastroenteritis (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 1 | 3 | 1 | 1 | 8
Nausea (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 5
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1 | 0 | 0 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1 | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0 | 0 | 5
Fatigue (General disorders) | 1 | 5 | 7 | 3 | 0 | 10
Pain (General disorders) | 2 | 1 | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 9 | 10 | 7 | 5 | 0 | 16
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 3
Helicobacter pylori (Investigations) | 0 | 0 | 3 | 2 | 3 | 3
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 2 | 1 | 1 | 0 | 0 | 3
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 3
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.